CLINICAL TRIAL: NCT06554509
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II/III Clinical Study of the Efficacy and Safety of SHR-1819 Injection in Adult Patients With Prurigo Nodularis
Brief Title: Clinical Study of the Efficacy and Safety of SHR-1819 Injection in Adult Patients With Prurigo Nodularis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1819-302
Record Dates: First submitted 2024-08-05; First posted 2024-08-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Prurigo Nodularis

STUDY DESIGN:
Intervention Model Description: SHR-1819 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A：SHR-1819 injection dose 1 (Experimental)
  Interventions: Drug: SHR-1819 injection
- Treatment group B：SHR-1819 injection dose 2 (Experimental)
  Interventions: Drug: SHR-1819 injection
- Treatment group C：SHR-1819 injection dose 3 (Experimental)
  Interventions: Drug: SHR-1819 injection
- Treatment group D：placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1819 injection — SHR-1819 injection
  Arms: Treatment group A：SHR-1819 injection dose 1; Treatment group B：SHR-1819 injection dose 2; Treatment group C：SHR-1819 injection dose 3
Drug: Placebo — placebo
  Arms: Treatment group D：placebo

SUMMARY:
This trial was designed to evaluate the efficacy and safety of SHR-1819 injection in patients with Prurigo Nodularis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign informed consent forms prior to the commencement of any proceedings related to the study, are able to communicate smoothly with the investigator, understand and are willing to complete the study in strict compliance with the requirements of this clinical research protocol.
2. The age was ≥18 at the time of signing the informed consent and gender is unlimited.
3. Have prurigo Nodularis at screening.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Major surgeries are planned for the duration of the study.
3. Has an active skin disease (such as chronic lichen simplex, psoriasis, chronic photosensitive dermatitis, etc.) or skin complications due to other diseases that may affect the evaluation of PN.
4. History of clinically significant diseases (e.g., circulatory system abnormalities, endocrine system abnormalities, neurological disorders, hematologic disorders, immune system disorders, psychiatric disorders, and metabolic instability) that the researcher believes that participation in the study poses a risk to the safety of the subject or that the disease/illness worsens during the study period will affect the effectiveness or safety analysis.
5. Treated with biologics targeting IL-4Rα (such as dupliumab), or participated in previous clinical studies of biologics targeting IL-4Rα, including SHR-1819 injection.
6. Screening for people with a history of heavy alcohol consumption or substance abuse in the 6 months prior to screening.
7. Diagnosis of moderate to severe AD during the screening/lead-in period or prior to randomization.
8. Subjects with malignancy prior to screening (except for squamous cell carcinoma of the skin, basal cell carcinoma, or carcinoma in situ of the cervix that are completely resected and have no evidence of recurrence).
9. Use of other biologics (such as omalizumab) within 3 months or 5 half-lives prior to screening, whichever is longer as confirmation.
10. Other conditions that, in the opinion of the investigator, are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Phase II: Proportion of subjects with a ≥4-point reduction from baseline in the weekly mean of the Most Intense Pruritus Numeric Rating Scale (WI-NRS) at Week 16 | up to 16 weeks
  Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity.
Phase III: Proportion of subjects with a ≥4-point reduction from baseline in the weekly mean of the Most Intense Pruritus Numeric Rating Scale (WI-NRS) at Week 24 | up to 24 weeks
  Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity.

SECONDARY OUTCOMES:
Phase II: Weekly mean change from baseline and percentage change in weeks 2, 4, 8, 12, and 16 of WI-NRS | up to 16 weeks
  Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity.
Phase II: Proportion of subjects with IGA CNPG-S score of 0/1 at weeks 4, 8, 12 and 16 | up to 16 weeks
  It consists of a 5-point scale ranging from 0 to 4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe PN.
Phase II: Change from baseline in Dermatology Life Quality Index (DLQI) score at weeks 4, 8, 12, 16 | up to 16 weeks
  It comprises of set of 10 questions. Responses to each question were assessed on a 4-point Likert scale ranged from 0 (not at all) to 3 (very much). Scores from all 10 questions added up to give total DLQI scores ranged from 0 (not at all) to 30 (very much), higher scores indicated more impact on quality of life.
Phase III: Proportion of subjects with an IGA CNPG-S score of 0/1 at week 24 | up to 24 weeks
  It consists of a 5-point scale ranging from 0 to 4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe PN.
Phase III: Proportion of subjects with IGA CNPG-S score of 0/1 at weeks 4, 8, 12, 16, and 20 | up to 24 weeks
  It consists of a 5-point scale ranging from 0 to 4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe PN.
Phase III: Change from baseline in Dermatology Life Quality Index (DLQI) score at weeks 4, 8, 12, 16, 20, 24 | up to 24 weeks
  It comprises of set of 10 questions. Responses to each question were assessed on a 4-point Likert scale ranged from 0 (not at all) to 3 (very much). Scores from all 10 questions added up to give total DLQI scores ranged from 0 (not at all) to 30 (very much), higher scores indicated more impact on quality of life.
Phase II/III: The concentration of SHR-1819 in serum: AUC | From the beginning of administration to the 24/32th week
  The concentration of SHR-1819 in plasma will be determined
Phase II/III: Changes in the level of IgE in the serum | From the beginning of administration to the 24/32th week
  Changes in the level of biomarkers in serum
Phase II/III: Immunogenic endpoint: evaluate the incidence of ADA positivity for SHR-1819 | From the beginning of administration to the 24/32th week
  Incidence of immunogenicity in the body

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided